CLINICAL TRIAL: NCT02168153
Title: Assessment of Chiropractic Treatment Using Reaction and Response Times in Members of the Special Operation Forces (ACT2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Palmer College of Chiropractic (Other); Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0352
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Physiological Measurements of Response and Reaction Times
Keywords: Chiropractic Manipulative Therapy; Reaction Times; Response Times; Special Forces; Biomechanical Assessments
MeSH Terms: interventions — Manipulation, Spinal; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chiropractic Manipulative Therapy (Active Comparator): Participants will complete questionnaires and biomechanical assessments, and additionally receive CMT treatment.
  Interventions: Other: Chiropractic Manipulative Therapy
- Wait-List Control Group (Placebo Comparator): Participants will complete questionnaires and biomechanical assessments
  Interventions: Other: Wait-list

INTERVENTIONS:
Other: Chiropractic Manipulative Therapy — Participants will receive chiropractic spinal manipulative therapy consisting of High velocity low amplitude (HVLA) spinal manipulative procedures. These procedures are typically associated with a quick manual thrust and a cavitation sound. For the cervical spine, a procedure called a cervical index pillar push, thoracic manipulation will occur with unilateral or bimanual contacts in the prone or supine positions and lumbar/pelvis manipulation will be performed with a procedure referred to as side-lying or side-posture.
  Other Names: Chiropractic Care; Spinal Manipulation
  Arms: Chiropractic Manipulative Therapy
Other: Wait-list — Participants randomized to the wait-list control group will complete questionnaires and perform the same study procedures as those randomized to the chiropractic manipulative therapy arm. After completing the required 2-week waiting period, those who wish to receive chiropractic manipulative therapy will be eligible to schedule treatment visits.
  Arms: Wait-List Control Group

SUMMARY:
This study is a randomized controlled trial designed to evaluate changes in reaction times (RTs) and response times (RespTs) following chiropractic treatment compared to controls in the Special Forces Qualified (SFQ) population, including Special Operation Forces who are part of the 160th SOAR regiment on flight status.

DETAILED DESCRIPTION:
The Assessment of Chiropractic Treatment 2 (ACT2) assesses changes in reaction/response times following Chiropractic Manipulative Therapy (CMT) using a randomized controlled trial in members of SFQ or SOAR. This population is faced with simultaneous physiological and cognitive demands. The ability to give an accurate and appropriate motor response in a short time is required for successful completion of the types of missions they are expected to undertake.

It is possible that chiropractic care can improve performance in reaction and response times in populations that have low back pain and in populations that are asymptomatic. One possible theory for improvement, even in asymptomatic persons, is that they may have experienced an insult or stress to the body which is subclinical but alters their ability to function in an optimal manner. Thus a person may be asymptomatic and able to accomplish many activities in a normal manner, but when stressed to the limits of maximum capability, the effects of subclinical abnormalities may cause that person to function at a less than optimal level. If CMT is able to restore normal, more efficient mechanisms of functioning, it is therefore possible that the performance of challenging tasks could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Age range at least 20 years of age
* Written informed consent
* Active duty SFQ personnel or Special Operation Forces who are part of the 160th SOAR regiment on flight status stationed at the Ft. Campbell, KY military site

Exclusion Criteria:

* Pain Intensity (NIH's PROMIS- question #29) > 4 at the Initial Visit
* Additional diagnostic procedure needed (e.g. x-ray)
* Bone and joint pathology contraindications for CMT. Potential participants with recent spinal fracture, concurrent spinal or paraspinal tumor(s), spinal or paraspinal infection(s), inflammatory arthropathies and significant osteoporosis will be referred for appropriate care.
* Other contraindications for CMT (i.e., unstable spinal segments, cauda equina syndrome)
* Currently being treated for traumatic brain injury (TBI)
* Reasonable chance that within 2-4 weeks of initial participation they may be unable to complete the study, i.e., deployment, receive orders for a distant duty assignment or training site or otherwise be absent from the current military site over the study participation period.
* Received care from a Doctor of Chiropractic within the past 30 days.
* Pregnant or planning to become pregnant within 4 weeks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Coulter, Ph.D, Principal Investigator — RAND
Locations (1):
- Blanchfield Army Community Hospital, Fort Campbell North, Kentucky, United States

REFERENCES:
- [Background] DeVocht JW, Smith DL, Long CR, Corber L, Kane B, Jones TM, Goertz CM. The effect of chiropractic treatment on the reaction and response times of special operation forces military personnel: study protocol for a randomized controlled trial. Trials. 2016 Sep 20;17(1):457. doi: 10.1186/s13063-016-1580-1. PMID 27645465
- [Background] DeVocht JW, Vining R, Smith DL, Long C, Jones T, Goertz C. Effect of chiropractic manipulative therapy on reaction time in special operations forces military personnel: a randomized controlled trial. Trials. 2019 Jan 3;20(1):5. doi: 10.1186/s13063-018-3133-2. PMID 30606225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were primarily referred to the project manager from physical therapists and other healthcare providers. The remainder of the participants were recruited from informational presentations by the site project manager, informational emails, and the SOF newsletter.
Period: Overall Study
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Started | 60 | 60
Completed | 57 | 60
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5.1) | 33.2 (6.1) | 33.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 60 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 2 | 5
  White | 54 | 55 | 109
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Simple Reaction Time With the Dominant Hand
Description: Handedness of the participants will be determined on the basis of self-report. The subject will react to the appearance of visual prompts on the screen by pressing a button with the thumb of their dominant hand. A set consists of 11 prompts shown in sequence with a time period between the response to one prompt and the appearance of the next prompt ranging from 0.5 to 4.0 seconds in random order. The outcome variable for this test, the mean reaction time, is the average of the length of time between the appearance of each prompt and the press of the button in response to that prompt.
Time Frame: Week 1-Study Visit 2, Week 2-Final Visit, Change from Visit 2 to Final Visit
Population: Missing data for the simple hand reaction tests are due to a technical problem in early data collection. Once identified, the problem was corrected. Because data collected before the technical issue was corrected were unreliable and likely inaccurate, they were not included in the analysis for this measure.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Number analyzed (Participants) | 37 | 40
millisecond (ms)
  Week 1-Study Visit 2 | 258.7 (48.6) | 254.7 (46.4)
  Week 2-Final Visit | 252.6 (33.7) | 252.3 (49.3)
  Change from Visit 2 to Final Visit | -4.88 (42.57) | -1.68 (53.56)
Statistical Analysis 1: Comparison: Chiropractic Manipulative Therapy vs Wait-List Control Group; Between group differences; Test type: Superiority; p = 0.76, ANCOVA; adjusted for age; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-25.75 to 18.77]

2. Primary Outcome: Simple Reaction Time With the Dominant Foot
Description: This test will be done in a manner similar to that for the dominant hand except that the participants will press a pedal with their dominant foot.
Time Frame: Week 1-Study Visit 2, Week 2-Final Visit, Change from Visit 2 to Final Visit
Population: Missing data for the simple foot reaction tests are due to a technical problem in early data collection. Once identified, the problem was corrected. Because data collected before the technical issue was corrected were unreliable and likely inaccurate, they were not included in the analysis for this measure.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Number analyzed (Participants) | 37 | 40
millisecond (ms)
  Week 1-Study Visit 2 | 291.9 (41.8) | 300.6 (41.8)
  Week 2-Final Visit | 300.6 (32.1) | 307.0 (49.3)
  Change from Visit 2 to Final Visit | 8.65 (39.98) | 7.88 (42.83)
Statistical Analysis 1: Comparison: Chiropractic Manipulative Therapy vs Wait-List Control Group; Between group differences; Test type: Superiority; p = 0.92, ANCOVA; adjusted for age; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-18.04 to 19.98]

3. Primary Outcome: Choice Reaction Time
Description: Prompts on the screen will occur with the same time interval (1 second) in between the press of a button or pedal in response to one prompt and the appearance of the next prompt. Each prompt could be for either hand or either foot and the position of the prompt on the computer screen will indicate which thumb or foot should be used. If the wrong button or pedal is pressed, the software still goes on to the next prompt, but keeps track of how many incorrect responses were made. A set consists of a sequence of 41 prompts. The outcome variable for this test, mean reaction time, is the average length of time between each prompt's appearance and the participant's response.
Time Frame: Week 1-Study Visit 2, Week 2-Final Visit, Change from Visit 2 to Final Visit
Population: 3 participants in the Chiropractic group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: Millisecond (ms)
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Number analyzed (Participants) | 57 | 60
Millisecond (ms)
  Week 1-Study Visit 2 | 426.1 (56.2) | 445.9 (72.9)
  Week 2-Final Visit | 421.7 (55.7) | 436.4 (67.9)
  Change from Visit 2 to Final Visit | -6.42 (44.06) | -9.51 (53.29)
Statistical Analysis 1: Comparison: Chiropractic Manipulative Therapy vs Wait-List Control Group; Between group differences; Test type: Superiority; p = 0.70, ANCOVA; adjusted for age; Mean Difference (Final Values) = 3.49, 95% CI 2-sided [-14.4 to 21.39]

4. Primary Outcome: Response Time Involving the Dominant Hand (Fitts Law Test)
Description: Participants perform a computerized simple target acquisition task (a Fitts Law task) to investigate their response times using a mouse with their dominant hand. The participant will complete a block, a series of target selections on a computer monitor, by working through 32 trials. That is, 32 pairs of 'hits' - meaning the mouse was clicked when the cursor was inside each of two circles that appear on the screen. The measured outcome from this task will be the sum of the times required to complete each trial.
Time Frame: Week 1-Study Visit 2, Week 2-Final Visit, Change from Visit 2 to Final Visit
Population: 3 participants in the Chiropractic group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Number analyzed (Participants) | 57 | 60
millisecond (ms)
  Week 1-Study Visit 2 | 65.9 (0.40) | 67.1 (0.66)
  Week 2-Final Visit | 66.3 (0.72) | 66.6 (0.32)
  Change from Visit 2 to Final Visit | 0.412 (3.710) | -0.548 (3.731)
Statistical Analysis 1: Comparison: Chiropractic Manipulative Therapy vs Wait-List Control Group; Between group differences; Test type: Superiority; p = 0.15, ANCOVA; adjusted for age; Mean Difference (Final Values) = 0.988, 95% CI 2-sided [-0.373 to 2.349]

5. Primary Outcome: Response Time Involving Whole Body Movement (T-wall)
Description: Participants will stand in front of the t-wall which is a commercially available device with a 4 x 8 foot bank of square buttons that are each 8 cm per side. When test is begun, one of the buttons lights up. The participant hits that button with either hand. The light inside that button then goes out and another button lights up until that one is hit. This process continues for a random sequence of 100 buttons. When last button is hit, all the buttons light up momentarily to indicate that the test is over. The measured outcome from this test is the time from when the first button is hit to when the last of the random sequence of 100 buttons is hit.
Time Frame: Week 1-Study Visit 2, Week 2-Final Visit, Change from Visit 2 to Final Visit
Population: 3 participants in the Chiropractic group were lost to follow-up.
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
Number analyzed (Participants) | 57 | 60
millisecond (ms)
  Week 1-Study Visit 2 | 49.1 (4.7) | 50.1 (4.2)
  Week 2-Final Visit | 47.2 (4.2) | 48.5 (4.4)
  Change from Visit 2 to Final Visit | -2.00 (2.40) | -1.59 (2.1)
Statistical Analysis 1: Comparison: Chiropractic Manipulative Therapy vs Wait-List Control Group; Between group differences; Test type: Superiority; p = 0.32, ANCOVA; adjusted for age; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.24 to 0.41]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were defined as any unexpected or unusual medical occurrence during the conduct of the trial that may or may not have a causal relationship with trial procedures.
Arm/Group | Chiropractic Manipulative Therapy | Wait-List Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No